CLINICAL TRIAL: NCT00031577
Title: A Phase I Study Of Taxol And Involved Field Radiation Therapy For Newly Diagnosed Intrinsic Gliomas Of Childhood
Brief Title: Paclitaxel Plus Radiation Therapy in Treating Children With Newly Diagnosed Brain Stem Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative closure 9/22/2006. Decline in enrollment at CHOP. due to competing protocols with new agents.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1999-6-1780; CHP-623; BMS-CHP-623; NCI-V01-1677; CDR0000069064
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2014-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Paclitaxel may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of combining paclitaxel with radiation therapy in treating children who have newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of paclitaxel when combined with involved-field radiotherapy in children with newly diagnosed, diffuse, intrinsic brain stem glioma.
* Determine the toxicity of this regimen in these patients.
* Assess the antitumor activity of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of paclitaxel.

Patients receive induction therapy comprising paclitaxel intravenously (IV) over 1 hour once weekly and involved-field radiotherapy (after paclitaxel infusion) once daily, 5 days a week, for 6 weeks.

Beginning 6 weeks after completion of induction therapy, patients may receive maintenance therapy comprising paclitaxel IV over 1 hour once every 3 weeks for a total of 8 courses. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 12 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, diffuse, intrinsic brain stem glioma by clinical examination and magnetic resonance imaging (MRI)

  * Histologic verification not required
  * Intrinsic (more than 50% intra-axial) involvement of the pons, pons and medulla, pons and midbrain, or entire brain stem allowed
  * Contiguous involvement of the thalamus or upper cervical cord allowed

PATIENT CHARACTERISTICS:

Age:

* 3 to 21 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin less than 1.5 times normal
* serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) less than 2.5 times normal

Renal:

* Creatinine less than 1.5 times normal

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use a highly effective method of contraception for female patients or barrier contraception for male patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No other concurrent anticancer chemotherapy

Endocrine therapy:

* Concurrent corticosteroid therapy for increased intracranial pressure allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent cytochrome P450-inducing anticonvulsants (e.g., phenytoin or carbamazepine) during paclitaxel therapy
* Other concurrent anticonvulsants (e.g., valproic acid) for pre-existing seizure disorder allowed

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 1999-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean B. Belasco, MD, Study Chair — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Winship Cancer Institute of Emory University, Egleston, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania